CLINICAL TRIAL: NCT04886739
Title: Safety and Effectiveness of CGB-400 Topical Gel for the Treatment of Inflammatory Lesions of Rosacea: A Randomized, Double-Blind, Vehicle-Controlled Proof of Concept Study
Brief Title: CGB-400 Topical Gel for the Treatment of Inflammatory Lesions of Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGB-400-002
Record Dates: First submitted 2021-04-30; First posted 2021-05-14 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CGB-400 Topical Gel (Experimental): Topical administration twice daily for 12 weeks
  Interventions: Drug: CGB-400
- Vehicle Gel (Placebo Comparator): Topical administration twice daily for 12 weeks
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: CGB-400 — Topical gel
  Arms: CGB-400 Topical Gel
Drug: Vehicle Gel — Topical gel
  Arms: Vehicle Gel

SUMMARY:
This is a multicenter, randomized, double-blind, vehicle-controlled, parallel design study evaluating the efficacy and safety of CGB-400 Topical Gel for the treatment of inflammatory lesions of rosacea. The study consists of a 12-week double-blind treatment period with clinic visits at Baseline (Day 0), and Weeks 2, 4, 8, and 12.

Approximately 80 subjects will be enrolled and randomized at a 1:1 ratio to treatment with either CGB-400 Topical Gel (40%) BID or Vehicle Gel BID.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative UPT at Baseline and practice a reliable method of contraception throughout the study.
* Clinical diagnosis of papulopustular facial rosacea.
* Investigator Global Assessment (IGA) score of 3 or 4 (i.e., moderate or severe).
* Facial inflammatory lesion count (i.e., papules and pustules) of ≥15 and ≤50 (excluding lesions involving the eyes and scalp) with ≤2 nodules.
* Willing to forego any other topical or non-topical treatment, cosmetic, OTC, or prescription on the study areas during treatment (other than sun protection or the study specified face wash and moisturizer).
* Willing to use the provided skincare regimen (e.g., face wash, moisturizer) during the study.
* In general good health as determined by medical history and physical examination at the time of screening (Investigator discretion).
* Sign the IRB-approved ICF (which includes HIPAA) prior to any study-related procedures being performed.

Exclusion Criteria:

* Female subjects that are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control (as specified in Section 5.1).
* Known hypersensitivity or previous allergic reaction to any constituent of the Investigational Product (i.e., essential oils, fragrance, choline, phosphatidylcholine, propylene glycol, limonene, cellulose).
* Any transient flushing syndrome.
* Particular forms of rosacea (ocular rosacea, rosacea conglobata, rosacea fulminans, isolated rhinophyma, granulomatous rosacea, phymatous rosacea, plaque-type rosacea lesions isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
* Papulopustular rosacea that had required systemic treatment within the past 12 months.
* Facial skin conditions that can interfere with reliable rosacea assessments (e.g., keloids, hypertrophic scarring, dense telangiectasia, plaque-like facial edema, recent facial surgery, etc.).
* Facial dermatoses that may be confounded with papulopustular rosacea (e.g., perioral dermatitis, facial keratosis pilaris, seborrheic dermatitis, acne fulminans, etc.).
* History or presence of a skin condition/disease that is located in the treatment area(s) and might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, psoriasis, significant actinic damage, vitiligo, open wounds, infection, etc.).
* Basal cell carcinoma within 6 months of Visit 1.
* Uncontrolled systemic disease.
* Foreseen unprotected and intense/excessive UV exposure during the course of the study.
* Use of prohibited concomitant medications/procedures, as specified below in Table 1, during the study or within the defined washout periods.
* Scheduled or planned surgical procedures during the course of the study.
* Unable or unwilling to comply with any of the study requirements.
* Medical or psychiatric conditions, or a personal situation, that may increase the risk associated with study participation or may interfere with interpretation of study results or subject compliance and, in the opinion of the PI, makes the subject inappropriate for study entry.
* Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
* Exposure to any other investigational drug/device within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Inflammatory Lesion Count | Week 12
  Numerical count of inflammatory lesions (pustules and papules)
Investigator Global Assessment (IGA) | Week 12
  * 0 - Clear; No inflammatory lesions present; at most mild erythema
  * 1 - Almost clear; Very mild erythema present. Very few small papules/pustules
  * 2 - Mild; Mild erythema. Several small papules/pustules
  * 3 - Moderate; Moderate erythema. Several small or large papules/pustules
  * 4 - Severe; Severe erythema. Numerous small and/or large papules/pustules

SECONDARY OUTCOMES:
Inflammatory Lesion Count | Weeks 2, 4, and 8
  Numerical count of inflammatory lesions (pustules and papules)
Investigator Global Assessment (IGA) | Weeks 2, 4, and 8
  * 0 - Clear; No inflammatory lesions present; at most mild erythema
  * 1 - Almost clear; Very mild erythema present. Very few small papules/pustules
  * 2 - Mild; Mild erythema. Several small papules/pustules
  * 3 - Moderate; Moderate erythema. Several small or large papules/pustules
  * 4 - Severe; Severe erythema. Numerous small and/or large papules/pustules
Rosacea Quality of Life (RosaQoL) Questionnaire | Week 12
  Patient Reported Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Cage Bio Investigative Site 1, Fremont, California, United States